CLINICAL TRIAL: NCT05341193
Title: PD-1 Inhibitor and Bevacizumab Replace Cisplatin in Induction, Concurrent, and/or Adjuvant Therapy for High-risk Locoregionally Advanced Nasopharyngeal Carcinoma.
Brief Title: PD-1 Blockade and Bevacizumab Replace Cisplatin in Locoregionally Advanced Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Ming-Yuan Chen, Chief physician, Proffessor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-CMY-2022-0416
Record Dates: First submitted 2022-04-18; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: antiangiogenesis; immunotherapy; Locoregionally Advanced Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Adjuvants, Pharmaceutic; Bevacizumab; toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low risk (Experimental): Patients will receive induction therapy with toripalimab plus bevacizumab and gemcitabine every 3 weeks for 3 cycles before radiotherapy, then followed by IMRT and concurrent therapy with toripalimab plus bevacizumab for 2 cycles, then followed by adjuvant therapy with toripalimab every 3 weeks for a maximum of 1 year after radiotherapy.
  Interventions: Drug: Bevacizumab+Toripalimab+gemcitabine, adjuvant with Toripalimab
- high risk (Experimental): Patients will receive induction therapy with toripalimab plus bevacizumab and gemcitabine every 3 weeks for 3 cycles before radiotherapy, then followed by IMRT and concurrent therapy with toripalimab plus bevacizumab for 2 cycles, then followed by adjuvant therapy with toripalimab and bevacizumab every 3 weeks for a maximum of 1 year after radiotherapy.
  Interventions: Drug: Bevacizumab+Toripalimab+gemcitabine, adjuvant with Bevacizumab and Toripalimab

INTERVENTIONS:
Drug: Bevacizumab+Toripalimab+gemcitabine, adjuvant with Bevacizumab and Toripalimab — Induction therapy:
  Toripalimab (240mg iv drip)+Bevacizumab (7.5mg/kg iv drip)+gemcitabine (1,000 mg/m2), every 3 weeks for 3 cycles before radiotherapy.
  Concurrent therapy:
  Toripalimab (240mg iv drip)+Bevacizumab (7.5mg/kg iv drip), every 3 weeks for 2 cycles during radiotherapy.
  Adjuvant therapy:
  Toripalimab (240mg iv drip)+Bevacizumab (7.5mg/kg iv drip), every 3 weeks for 1 year after radiotherapy.
  Radiation:
  Intensity-modulated radiotherapy.
  Arms: high risk
Drug: Bevacizumab+Toripalimab+gemcitabine, adjuvant with Toripalimab — Induction therapy:
  Toripalimab (240mg iv drip)+Bevacizumab (7.5mg/kg iv drip)+gemcitabine (1,000 mg/m2), every 3 weeks for 3 cycles before radiotherapy.
  Concurrent therapy:
  Toripalimab (240mg iv drip)+Bevacizumab (7.5mg/kg iv drip), every 3 weeks for 2 cycles during radiotherapy.
  Adjuvant therapy:
  Toripalimab (240mg iv drip), every 3 weeks for 1 year after radiotherapy.
  Radiation:
  Intensity-modulated radiotherapy.
  Arms: low risk

SUMMARY:
At present, the treatment regimen of locally advanced nasopharyngeal carcinoma still needs to be further improved, and the focus of improvement lies in "replacing cisplatin with high-efficiency and low-toxicity treatment regimen". Considering the synergistic effect among radiotherapy, immunotherapy and anti-angiogenesis therapy, we chose PD-1 inhibitor combined with bevacizumab to replace cisplatin chemotherapy.

DETAILED DESCRIPTION:
We plan to use PD-1 inhibitor combined with bevacizumab to replace cisplatin (induction + concurrent ± adjuvant) in patients with locally advanced nasopharyngeal carcinoma. Considering the safety of the original study, we will set up two groups for the adjuvant treatment stage: one group will only use PD-1 inhibitor at the adjuvant treatment stage (low risk group), and the other group will use bevacizumab +PD-1 inhibitor combined treatment (high risk group). Once the efficacy and safety of this protocol are confirmed, it may provide a new treatment option for locally advanced nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation with Written informed consent.
2. Age ≥ 18 years and ≤ 65 years.
3. Histologically confirmed with Nonkeratinizing carcinoma of the nasopharynx (differentiated or undifferentiated type).
4. Original clinical staged as III-IVa (according to the 8th AJCC edition).
5. Stage III patients should meet the criteria of EBV DNA≥4000 cps/ml.
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1.
7. Patients must have adequate organ function:

   1. White blood cell count (WBC)≥4.0×109 /L, Hemoglobin ≥ 90g/L, Platelet count ≥100×109/L.
   2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×upper limit of normal (ULN),serum total bilirubin (TBIL) ≤2.0 times the upper limit of normal (ULN) .
   3. Adequate renal function: creatinine clearance rate≥60 ml/min or Creatinine ≤1.5× upper limit of normal value.
   4. INR, APTT≤1.5 x ULN.

Exclusion Criteria:

1. Subjects with recurrent or metastatic nasopharyngeal carcinoma.
2. Histologically or cytologically confirmed with keratinizing squamous cell carcinoma of the nasopharynx.
3. Prior therapy with systemic therapy for nasopharyngeal carcinoma.
4. Prior exposure to immune checkpoint inhibitors,including anti-PD-1, anti-PD-L1, anti-CTLA-4 antibodies.
5. Prior exposure to antiangiogenic agents.
6. Tumor invasion to the intracranial with clinical symptoms accompanied by cerebral edema, requiring hormone therapy.
7. Any grade ≥2 bleeding event (according to CTCAE 5.0) occurred within 4 weeks prior to enrollment.
8. Subjects with an active, known or suspected autoimmune disease.
9. Subjects with clinically significant cardiovascular and cerebrovascular diseases.
10. Subjects with high blood pressure who cannot be controlled well with antihypertensive drugs.
11. Subjects with previous digestive tract bleeding history within 3 months or evident gastrointestinal bleeding tendency.
12. Subjects with arterial / venous thrombosis events occurred within 6 months of the first dose.
13. Women in the period of pregnancy, lactation, or reproductive without effective contraceptive measures.
14. Seropositivity for human immunodeficiency virus (HIV).
15. Known history of other malignancies (except cured basal cell carcinoma or carcinoma in situ of the cervix).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-04-30 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
grade ≥3 nasopharyngeal necrosis or hemorrhage | At the end of each cycle (each cycle is 21 days)
  Incidence of nasopharyngeal necrosis or massive hemorrhage (grade ≥3).
  Grade ≥3 hemorrhage: Grade 3, Transfusion indicated; invasive intervention indicated; hospitalization. Grade 4, Life-threatening consequences; urgent intervention indicated (e.g., tracheotomy or intubation). Grade 5, death.
  Grade ≥3 nasopharyngeal necrosis: Grade 3, Severe pain; unable to adequately aliment or hydrate orally; limiting self care ADL. Grade 4, Life-threatening consequences; urgent intervention indicated.
  Grade 5, death.

SECONDARY OUTCOMES:
Objective response rate | 3 weeks after indution therapy; 3 months after concurrent therapy
  The proportion of patients whose tumors shrink to a certain size and maintain such size for a certain period of time, including patients with complete response (CR) and partial response (PR).
Progression-free survival | 3 year
  Progress-free survival is calculated from the date of enrollment to the date of the first progression at any site or death from any cause or censored at the date of the last follow-up.
Overall survival | 3 year
  Overall survival is calculated from the date of enrollment to the date of the death from any cause or censored at the date of the last follow-up.
Locoregional failure-free survival (LRRFS) | 3 year
  Defined as the time from registration to local or regional relapse, or death from any cause.
Distant metastasis-free survival (DMFS) | 3 year
  Defined as the time from registration to distant metastasis, or death from any cause.
Incidence rate of adverse events (AEs) | 3 year
  Analysis of acute and late adverse events (AEs) are evaluated. Numbers of patients of treatment-related adverse events (acute toxicity) and late radiation toxicities were assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-yuan Chen, MD, PhD, Study Chair — Sun Yat-sen University
Locations (1):
- Department of Nasopharyngeal Carcinoma, Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China